CLINICAL TRIAL: NCT03508648
Title: Phase 2 Durability Extension Study to Assess Clinical Activity and Safety of Enobosarm (GTx-024) in Postmenopausal Women With Stress Urinary Incontinence
Brief Title: Durability Extension Study to Assess Clinical Activity and Safety of Enobosarm (GTx-024) in Stress Urinary Incontinence
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy from primary study
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: G201003
Record Dates: First submitted 2018-04-16; First posted 2018-04-26 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — ostarine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Matching Placebo (Placebo Comparator): Subjects previously enrolled in the placebo arm of study G201002.
  Interventions: Drug: Matching Placebo
- 1 mg GTx-024 (Active Comparator): Subjects previously enrolled in the 1 mg GTx-024 arm of study G201002.
  Interventions: Drug: GTx-024
- 3 mg GTx-024 (Active Comparator): Subjects previously enrolled in the 3 mg GTx-024 arm of study G201002.
  Interventions: Drug: GTx-024

INTERVENTIONS:
Drug: GTx-024 — Subjects will not be provided with any study treatments and will be off-drug during this extension study. Intervention was administered during study G201002.
  Other Names: enobosarm
  Arms: 1 mg GTx-024; 3 mg GTx-024
Drug: Matching Placebo — Subjects will not be provided with any study treatments and will be off-drug during this extension study. Intervention was administered during study G201002.
  Arms: Matching Placebo

SUMMARY:
The study will enroll only from the first 225 subjects who were randomly assigned to treatment in G201002 (irrespective of the treatment allocation, i.e., GTx-024 or placebo) and who have completed the 12-week treatment period and 16-week durability period to assess the long-term durability of response to GTx-024 on SUI symptoms. The extension study will follow subjects for an additional 20 weeks to help better assess the durability of response in these subjects and will provide additional efficacy and safety data for the subjects. Subjects will not be provided with any study treatments and will be off-drug during this extension study.

ELIGIBILITY:
Inclusion Criteria:

* Be one of the first 225 subjects who were randomly assigned to treatment in G201002 (Phase 2 study) and have completed the 12-week treatment and 16-week durability periods
* Be able to read, understand, and provide written, dated informed consent prior to enrollment in the current study (within 2 weeks of completing G201002) and be likely to comply with the study protocol and communicate with study personnel about AEs and other clinically important information
* Agree to maintain a stable dose of any medication known to affect lower urinary tract function, including but not limited to anticholinergics, tricyclic antidepressants, beta-3 adrenergic agonists, or α-adrenergic blockers, throughout the duration of the study

Exclusion Criteria:

* Starts any new treatment (medication, pelvic floor physical therapy, or other treatment known to impact the pelvic floor) after completing G201002 that is known or suspected to affect lower urinary tract function, including vaginal rejuvenation
* Has a current or past history of any physical condition that, in the investigator's opinion, might put the subject at risk or interfere with interpretation of study results

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Durability of Response, stress incontinence | baseline to 20 weeks
  Change from G201002 baseline in the mean number of stress incontinence episodes per day
Durability of Response, patient global impression of severity | baseline to 20 weeks
  Change from G201002 baseline in patient global impression of severity scale (PGI-S; scale: 1-normal, 2-mild, 3-moderate, 4-severe; representing severity of urinary tract dysfunction)
Durability of Response, patient global impression of improvement | baseline to 20 weeks
  Change from G201002 baseline in patient global impression of improvement scale (PGI-I; scale: 1-very much better, 2-much better, 3-a little better, 4-no change, 5-a little worse, 6-much worse, 7-very much worse; representing change in urinary tract dysfunction from initiation of therapy)

SECONDARY OUTCOMES:
Durability of Response, urge incontinence | baseline to 20 weeks
  Change from G201002 baseline in the mean number of urge incontinence episodes per day
Durability of Response, total incontinence | baseline to 20 weeks
  Change from G201002 baseline in the mean number of total (stress + urge) incontinence episodes per day

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Professor & Chair, Department of Urology, Oakland University Wm. Beaumont School of Medicine
Locations (46):
- United States (46):
  - Urology Center of Alabama, Homewood, Alabama
  - Coastal Clinical Research Inc, Mobile, Alabama
  - Alaska Clinical Research Center, Anchorage, Alaska
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Urology Associates Research, Englewood, Colorado
  - Women's Health Specialty Care, Farmington, Connecticut
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Tampa Bay Medical Research Inc, Clearwater, Florida
  - Midland Florida Clinical Research Center LLC, DeLand, Florida
  - Medical Research of Florida, Miami, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Mount Vernon Clinical Research LLC, Sandy Springs, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Idaho Urologic Institue, Meridian, Idaho
  - First Urology PSC, Jeffersonville, Indiana
  - Iowa Clinic, West Des Moines, Iowa
  - DelRicht Clinical Research, LLC, New Orleans, Louisiana
  - Regional Urology, Shreveport, Louisiana
  - Chesapeake Urology Associates PA, Hanover, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Bay State Clinical Trials, Watertown, Massachusetts
  - Beyer Research, Kalamazoo, Michigan
  - William Beaumont Hospital Urology Research, Royal Oak, Michigan
  - Women's Clinic of Lincoln, Lincoln, Nebraska
  - Sheldon J Freedman MD Ltd, Las Vegas, Nevada
  - Premier Urology Group, LL, Edison, New Jersey
  - Lawrence Obs Gyn clinical Research, Lawrenceville, New Jersey
  - Delaware Valley Urology, Mount Laurel, New Jersey
  - Accumed Research Associates, Garden City, New York
  - Manhattan Medical Research Practice PLLC, New York, New York
  - Circuit Clinical, West Seneca, New York
  - American Health Research Inc, Charlotte, North Carolina
  - Eastern Carolina Women's, New Bern, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Aventiv Research, Columbus, Ohio
  - Institute for Female Pelvic Medicine, Allentown, Pennsylvania
  - Urologic Consultants of Southeastern PA LLP, Bala-Cynwyd, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - Elligo - Austin Area OBGYN, Austin, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - Urology San Antonio Research PA, San Antonio, Texas
  - Synexus Clinical Research Advantage, Inc. - Wasatch Peak Family Practice, Layton, Utah
  - Seattle Womens: Health, Research, Gynocology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2015-08-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT03508648/Prot_000.pdf